CLINICAL TRIAL: NCT05782309
Title: Healthy Aging Through Dietary Intervention: Multiparametric Quantification of Function and Pathophysiology of the Aging Heart and Prevention of Age-associated Decline in Exercise Capacity Through Dietary Flavanols
Brief Title: Healthy Aging Through Dietary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AgingEx
Record Dates: First submitted 2023-02-09; First posted 2023-03-23 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Aging, Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flavanol (Experimental): 500 mg of flavanols twice daily
  Interventions: Drug: Flavanol
- Placebo (Placebo Comparator): nutrient matched control capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Flavanol — Assessement, supplementation for 30 days with either Placebo or Flavanols, Re-assessment
  Arms: Flavanol
Drug: Placebo — Assessement, supplementation placebo for 30 days with either Placebo or Flavanols, Re-assessment
  Arms: Placebo

SUMMARY:
To test the impact of flavanol supplementation of cardiac and vascular function and subsequently on exercise capacity in elderly individuals

ELIGIBILITY:
Inclusion Criteria:

* age 50-79

Exclusion Criteria:

* non-cardiac limitations of exercise capacity such as orthopedic or neurological disorders, BMI >35 kg/m2, active smoking, uncontrolled blood pressure, diabetes, COPD, atrial fibrillation, cardiomyopathy, coronary heart disease, valvular heart disease, cardiac pacemaker, acute respiratory tract infections, missing ability or missing cooperation to participate in the study

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | 30 days
  maximum power output during cardiopulmonary exercise testing
peakVO2 | 30 days
  maximum oxygen uptake during cardiopulmonary exercise testing

SECONDARY OUTCOMES:
flow mediated vasodilation (FMD) | 30 days
  marker for vascular function
Oxygen pulse | 30 days
  oxygen uptake per heart beat (VO2/HR) as measured during cardiopulmonary exercise testing
aortic stiffness | 30 days
  cardiac magnetic resonance assessment of aortic diameter, distensibility and flow
diastolic strain | 30 days
  cardiac magnetic resonance (CMR) based assessment of left ventricular strain
Left ventricular function | 30 days
  systolic ejection fraction calculated based on magnetic resonance volumetric assessment of left ventricle
left atrial volume index (LAVi) | 30 days
  cardiac magnetic resonance based assessment of left atrial volume index
brain natriuretic peptide (nt-proBNP) | 30 days
  blood chemistry, nt-proBNP measurement
aortic pulse wave velocity (PWV) | 30 days
  cardiac magnetic resonance based assessment of pulse wave velocity in ascending and descending aorta
diastolic strain rate (SR) | 30 days
  cardiac magnetic resonance (CMR) based assessment of left ventricular strain rate early and during atrial contraction

CONTACTS AND LOCATIONS:
Locations (1):
- Heinrich Heine University, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duse DA, Grone M, Ophoff N, Kramser N, Schweers H, Ottaviani J, Schroeter H, Quast C, Bonner F, Heiss C, Sansone R, Jung C, Kelm M, Erkens R. Cocoa flavanols alleviate early diastolic dysfunction by decreasing left atrial volume in a randomized double blinded trial in healthy older individuals. Food Funct. 2025 Nov 10;16(22):8836-8845. doi: 10.1039/d5fo02589c. PMID 41143317